CLINICAL TRIAL: NCT00207402
Title: A Pilot Trial of Combination Therapy With Interferon Alfacon1, Ribavirin, & Rosiglitazone in a Group of Insulin Resistant, Chronic Hepatitis C, GT 1 Patients Who Are Previous Relapsers or Nonresponders to Pegylated Interferon and Ribavirin
Brief Title: Infergen, Ribavirin & Avandia in Previous Relapsers or Nonresponders to Pegylated Interferon and Ribavirin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: InterMune (Industry)
Responsible Party: Principal Investigator, Stephen A Harrison, Principal Investigator, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2005.143
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Insulin resistance
MeSH Terms: conditions — Hepatitis C; Insulin Resistance | interventions — Rosiglitazone; interferon alfacon-1; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rosiglitazone (Active Comparator): Treatment with rosiglitazone 4 mg twice a day for 3 months prior to and during the course of 48 weeks of treatment with interferon alfacon-1 15mcg/0.5ml SQ daily and weight-based ribavirin.
  Interventions: Drug: rosiglitazone
- No Avandia (No Intervention): Monitoring period without rosiglitazone for 3 months prior to 48 weeks of interferon alfacon-1 15mcg/0.5ml SQ daily and weight-based ribavirin

INTERVENTIONS:
Drug: rosiglitazone — Infergen 15mcg/ d Avandia qd Ribavirin bid
  Other Names: Infergen (interferon alfacon-1); Avandia (rosiglitazone); Ribavirin
  Arms: rosiglitazone

SUMMARY:
Genotype 1 hepatitis C virus (HCV) patients who did not respond (did not lose virus during treatment) or relapsed (virus went away on treatment but came back after treatment was stopped) after treatment with at least twelve weeks of a pegylated (long-acting) interferon and ribavirin will be considered for this study. There are two purposes to this study: first, to determine how rosiglitazone, a medicine used to treat diabetes, affects the HCV viral load; and second, to determine if treatment of insulin resistance with rosiglitazone prior to therapy for HCV will improve sustained virologic response (loss of virus that continues beyond six months after completion of HCV therapy) to HCV therapy.

DETAILED DESCRIPTION:
This study will demonstrate the efficacy of treating insulin resistance with rosiglitazone in CHC, genotype 1 patients who have failed previous treatment with pegylated interferon and ribavirin. Pre-treatment with rosiglitazone may become the new standard of care prior to HCV therapy for those patients who are insulin resistant, increasing their chance for achieving an SVR on interferon alfacon-1 combination therapy and decreasing the morbidity and mortality associated with chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to give written informed consent and able to adhere to dose and visit schedules.
* Adult participants 18 years of age or older of either gender or any race. Participants who are over 65 years of age must be in generally good health.
* HCV-antibody (Ab) or HCV-RNA positive by polymerase chain reaction (PCR) for at least 6 months.
* Serum positive for HCV-RNA by PCR assay.
* Subjects must be previous nonresponders or relapsers on pegylated interferon and ribavirin therapy.
* Liver biopsy within 24 months prior to enrollment into the protocol.
* Compensated liver disease with the following minimum hematological, biochemical, and serologic criteria at the Screening Visit (WNL = within normal limits):

  * Hemoglobin values of < 12 gm/dL for females and < 13 gm/dL for males.
  * White blood cells (WBC) < 3,000/mm3
  * Neutrophil count < 1,500/mm3
  * Platelets < 65,000/mm3
  * Direct bilirubin, within 20% of upper limits of normal (ULN)
  * Indirect bilirubin, (WNL) (unless non-hepatitis related factors such as Gilbert's disease explain an indirect bilirubin rise. In such cases indirect bilirubin must be < 3.0 mg/dL [< 51.3 µmol/L]).
  * Albumin > 3 gm/dL
  * Serum creatinine < 20% of ULN
  * Thyroid stimulating hormone (TSH) WNL
  * Alpha fetoprotein value < 100 ng/mL.
* Reconfirmation and documentation that sexually active female subjects of childbearing potential are practicing adequate contraception during the treatment period and for 6 months following the last dose of study medication. Female subjects must not be breast-feeding.
* Reconfirmation that sexually active male subjects are practicing two acceptable methods of contraception during the treatment period and for 6 months following the last dose of study medication.

Exclusion Criteria:

* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Participants on insulin are excluded.
* Participants on metformin or another thiazolidinedione must have a three-month wash-out period to be considered for the study.
* Women who are pregnant or breast-feeding
* Males whose female partner is pregnant
* No other thiazolidinedione after liver biopsy and/or during the entire study (other than those subjects randomized to receive rosiglitazone during the study)
* Hepatitis C of non-genotype 1
* Suspected hypersensitivity to interferon, ribavirin, or rosiglitazone
* Any cause for liver disease other than chronic hepatitis C, insulin resistance, or non-alcoholic fatty liver disease (NAFLD), including but not limited to:

  * Hemochromatosis
  * Alpha-1 antitrypsin deficiency
  * Co-infection with hepatitis B virus (HBV) [serum hepatitis B surface antigen (HBsAg) positive]
  * Wilson's disease
  * Autoimmune hepatitis
  * Alcoholic liver disease (consumption of greater than 2 drinks a day on average)
  * Drug-related liver disease
* Any condition that would prevent the subject from having a liver biopsy.
* Hemoglobinopathies that could potentially compromise patient safety (e.g., beta thalassemia major, sickle cell disease)
* Evidence of advanced liver disease
* Participants with organ transplants other than cornea and hair transplant
* Any known preexisting medical condition that could interfere with the subject's participation in and completion of the protocol such as:

  * Preexisting psychiatric condition, especially severe depression, or a history of severe psychiatric disorder, such as major psychoses, suicidal ideation and/or suicidal attempt.
  * Participants with a history of mild depression may be considered for entry into the protocol provided that a pretreatment assessment of the subject's mental status supports that the participant is clinically stable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-10; Primary Completion 2010-01 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
There is change in viral kinetics with improvement of insulin sensitivity | 104 days

SECONDARY OUTCOMES:
There is significant improvement in the SVR obtained when treating insulin resistant patients with the insulin sensitizing medication, Avandia, prior to and during treatment with Infergen and ribavirin when compared to Infergen | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Harrison, MD, Principal Investigator — Brooke Army Medical Center; Shane Mills, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States